CLINICAL TRIAL: NCT03573167
Title: Mobile Phone-Based Motivational Interviewing to Reduce Alcohol Use Problems in Kenya
Brief Title: Mobile Phone-Based Motivational Interviewing in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Africa Institute of Mental and Brain Health (AFRIMEB) (Other)
Responsible Party: Principal Investigator, Valerie Harder, Associate Professor, University of Vermont
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CHRBSS 14-188
Record Dates: First submitted 2018-06-01; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-Person Motivational Interviewing (Active Comparator): In-Person Motivational Interviewing (MI) is the standard form of MI treatment delivered in person face to face at the primary care office. MI is a type of brief intervention that uses open-ended questions, affirmations, reflective listening, and summarizing as key tools and has been shown to treat a range of problem behaviors, including alcohol use disorders, by helping participants to identify and address ambivalence towards changing the behavior. MI is delivered in a communicative style that promotes individual autonomy and improves self-efficacy. The investigator provides counseling in-person with the participant for one session of MI lasting approximately 30 minutes.
  Interventions: Behavioral: In-Person Motivational Interviewing (MI)
- Mobile MI (Experimental): Mobile Motivational Interviewing (MI) is delivered by a counselor over the mobile phone, rather than in-person (face-to-face). MI is a type of brief intervention that uses open-ended questions, affirmations, reflective listening, and summarizing as key tools and has been shown to treat a range of problem behaviors, including alcohol use disorders, by helping the patient to identify and address ambivalence towards changing the behavior. MI is delivered in a communicative style that promotes individual autonomy and improves self-efficacy. The investigator provides counseling over the mobile phone with the participant for one session of mobile MI lasting approximately 30 minutes.
  Interventions: Behavioral: Mobile Motivational Interviewing (MI)
- Waitlist Control (No Intervention): After consenting to participate in the study, the Waitlist control participants receive no intervention for one (1) month, and then the Waitlist control participants are contacted by the investigators for follow up..

INTERVENTIONS:
Behavioral: In-Person Motivational Interviewing (MI) — This is a counseling intervention to support behavior change conducted in-person (face-to-face) between the investigator and the participant.
  Arms: In-Person Motivational Interviewing
Behavioral: Mobile Motivational Interviewing (MI) — This is a counseling intervention to support behavior change conducted entirely over the mobile phone between the investigator and the participant
  Arms: Mobile MI

SUMMARY:
The primary objective of this study was to test whether motivational interviewing (MI) provided over the mobile phone would reduce alcohol use among adults, including people living with HIV/AIDS, visiting primary care in Kenya. Heavy alcohol users voluntarily consented to being randomized to one of three study arms: standard in-person MI, mobile MI, or waitlist control receiving no intervention for 1 month followed by mobile MI. Alcohol use problems were assessed using validated screeners and changes in alcohol use were assessed at 1 month and 6 months after receiving the intervention. The investigators hypothesized that alcohol use would reduce after MI treatment compared to waitlist control, there would be no difference between standard in-person MI and mobile MI, and these reductions would be sustained out to six months following the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults visiting the primary care clinic and screening positive for potential alcohol use problems.

Exclusion Criteria:

* Persons younger than 18 years old, with severe psychiatric morbidity, or cognitive impairment were not eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction in alcohol use score as measured by the Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) from baseline to one (1) month. | 1 month
  The investigators compared the change in AUDIT-C alcohol use score from baseline to one (1) month after the intervention between the investigators' three study arms.
Reduction in alcohol use score as measured by the Alcohol Use Disorders Identification Test (AUDIT) and AUDIT-C from baseline to six (6) months. | 6 months
  The investigators compared the change in AUDIT and AUDIT-C alcohol use scores from baseline to six (6) months after the intervention between the investigators' two active study arms: 1) In-Person Motivational Interviewing (MI) and 2) Mobile MI.

SECONDARY OUTCOMES:
Reduction in alcohol use score as measured by the AUDIT and AUDIT-C moderated by HIV co-morbidity from baseline to one (1) month and from baseline to six (6) months. | 1 and 6 months
  The investigators compared the change in AUDIT and AUDIT-C alcohol use scores over time moderated by HIV status.
Reduction in alcohol use score as measured by the AUDIT moderated by mental health co-morbidity, as measured by the Achenbach System of Empirically Based Assessments (ASEBA) Adults Self-Report, from baseline to six (6) months. | 6 months
  The investigators compared the change in AUDIT alcohol use scores over time moderated by ASEBA mental health diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Harder, PhD, Principal Investigator — University of Vermont

IPD SHARING:
Plan to Share IPD: No